CLINICAL TRIAL: NCT02907983
Title: Stellate Ganglion Blockade for the Management of Vasomotor Symptoms
Brief Title: Stellate Ganglion Blockade in Post-Menopausal Women
Acronym: R01
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Audit panel terminated IRB approval and closed the study study.
Sponsor: Northwestern University (Other)
Collaborators: University of Illinois at Chicago (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00203490
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hot Flashes; Hot Flushes; Vasomotor Symptoms
Keywords: Menopause; Post-menopausal
MeSH Terms: conditions — Hot Flashes | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivicaine (Active Comparator): Stellate Ganglion Block injection with bupivicaine
  Interventions: Drug: Stellate Ganglion Block Injection with Bupivicaine
- Saline (Sham Comparator): Saline injection
  Interventions: Drug: Saline injection

INTERVENTIONS:
Drug: Stellate Ganglion Block Injection with Bupivicaine — A computer-generated stratified randomization scheme by self-reported race and by etiology of menopause (natural versus surgical menopause) will be used to assign participants to receive either a SGB with bupivacaine or a sham injection with saline. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card.
  Other Names: Marcaine
  Arms: Bupivicaine
Drug: Saline injection — A computer-generated stratified randomization scheme by self-reported race and by etiology of menopause (natural versus surgical menopause) will be used to assign participants to receive either a SGB with bupivacaine or a sham injection with saline. Randomization will be performed by the injectionist immediately before the injection procedure by opening an opaque envelope to reveal the participant number and group assignment printed on an index card.
  Other Names: Sodium chloride solution
  Arms: Saline

SUMMARY:
Hot flashes and night sweats (vasomotor symptoms, VMS) affect 80% of women during the menopausal transition (MT). VMS are associated with decreased quality of life, increased depressive and anxiety symptoms, memory complaints, sleep disturbance, and reduced work productivity. Hormone therapy (HT) is highly effective in reducing VMS, but the use of HT declined 75% to 80% in the U.S. after the Women's Health Initiative (WHI) raised safety concerns about HT. In 2013, the Food and Drug Administration (FDA) approved paroxetine, a selective serotonin reuptake inhibitor (SSRI; 7.5 mg), as the first non-hormonal treatment for VMS. SSRIs are an important treatment option for many women, but their use in treating VMS is limited by lower effectiveness when compared to HT, side effects, and relapse of symptoms following treatment discontinuation. Identifying safe and effective non-hormonal treatments for VMS remains a priority in women's health research.

Stellate ganglion blockade (SGB), used for decades in pain management, is a potential new approach to VMS treatment. Located in the cervical spine region, the stellate ganglia are part of the sympathetic nervous system. Although SGB is commonly performed to treat neuropathic pain, hyperhidrosis or vascular insufficiency, anatomic studies reveal connections between this ganglion and thermoregulatory regions of the brain, specifically the insular cortex.

In this clinical trial, we aim to assess whether stellate ganglion block (SGB) with bupivacaine, a local anesthetic, is an effective and safe non-hormonal intervention for women seeking relief from vasomotor symptoms (VMS), and identify the physiologic mechanisms underlying SGB effects. Outcomes will include frequency and intensity of hot flashes, objectively-measured VMS, mood, quality of life, sleep, and memory performance in 160 postmenopausal women with 50 or more moderate to very severe hot flashes per week as measured by self-report for six months. They will be reassessed at 3 and 6 months following the SGB or a sham intervention for objective hot flashes and quality of life measures. Mechanistic outcomes (neuroimaging) will be obtained at baseline and 3 months following the intervention. Ambulatory monitoring of sympathetic nervous system function (SKNA) will be performed at baseline before the procedure, during the procedure and 1 hour following the procedure. This will be repeated at 2 and four weeks following the SGB or sham procedure for 1 hour recordings.

DETAILED DESCRIPTION:
Scope:

Post-menopausal women with moderate to severe VMS will be enrolled as participants in this study.

Specific Goals and Objectives:

Primary Objective

1. To determine the effect of SGB for reducing frequency and intensity of menopausal VMS.

   Hypothesis 1a. Seven-day mean frequency of VMS will be lower in women randomized to active SGB compared to sham control.

   Hypothesis 1b. Seven-day mean intensity of VMS will be lower in women randomized to active SGB compared to sham control.

   Hypothesis 1c. The VMS Intensity (Frequency*Severity), will be lower in women randomized to active SGB compared to sham control.

   Secondary Objectives
2. To evaluate the effect of SGB on VMS Intensity, objective VMS, mood, memory, and sleep quality.

   Hypothesis 2a The frequency of objectively measured VMS will be lower in women randomized to active SGB compared to sham control.

   Hypothesis 2b. Depressive symptoms and memory, but not sleep quality, will improve more in women randomized to active SGB compared to sham control.

   Hypothesis 2c. The magnitude of improvements in memory will relate to the magnitude of reduction in VMS, even after controlling for sleep.
3. To probe the mechanisms by which SGB improves VMS.

Hypothesis 3a. In a nested sub study, neuroimaging assessments will reveal that compared to sham control, active SGB is associated with a) decreased functional connectivity in the default mode network during the resting state, particularly for networks supporting the insula and hippocampus; b) reduced activation in the hippocampus, dorsolateral prefrontal cortex, and anterior cingulate during a verbal memory task; and c) reduced activation in the amygdala during an emotion processing task.

Hypothesis 3b. Compared to sham control, SGB will immediately diminish ipsilateral stellate ganglion nerve activity and sympathetic tone as measured by skin sympathetic nerve monitoring (SKNA) and these effects will be reassessed at 2 and 4 weeks after the intervention to assess if effects of SGB on stellate ganglion activity are long lasting.

ELIGIBILITY:
Inclusion Criteria:

1. post-menopausal woman defined according to the following criteria: 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels ≥ 40 IU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
2. aged 40 to 70 years
3. 50 or more reported moderate-to-severe hot flashes per week
4. a minimum of two weeks of VMS diary recording prior to SGB
5. post-menopausal women whose vasomotor symptoms are refractory to approved oral treatments (i.e., hormone therapy or paroxetine) or for whom hormone therapy is contraindicated or for women who refuse any oral therapy
6. willingness to undergo fluoroscopy-guided SGB or sham treatment.
7. safety labs within 30 days of SGB intervention

Exclusion Criteria:

1. conditions that preclude SGB or sham intervention (e.g., anatomic abnormalities of the anterior neck or cervical spine ; goiter, cardiac/pulmonary compromise; contralateral (left-sided) phrenic nerve paralysis or diaphragmatic paresis; history of seizure, coma, or stroke; history of neurologic deficit to the brachial plexus or an abnormal brachial plexus neurologic exam; history of Zenker's diverticulum; acute illness/infection; coagulopathy or bleeding abnormalities; INR >1.3; hemoglobin<9.0, platelets <100,000, BUN ≥ 30mg/dl; creatinine ≥ 2 mg/ml; ALT (SGPT), AST (SGOT), Alk Phos ≥ three times the upper limit of normal; serum potassium (K+) ≤ 3.5 or ≥ 5.0 mEq/L allergic reactions or contraindications to a local anesthetic or contrast dye, systolic blood pressure (SBP) >140 mm Hg or diastolic blood pressure (DBP) >90 mm Hg, pregnancy
2. If LMP is between 6 to 12 months, FSH < 40
3. use of treatments less than the washout period and throughout study participation that can affect VMS frequency or severity, including oral (2 months) or transdermal hormone therapy(1 month), botanicals (e.g., soy, red clover, black cohosh, etc.)(1 month), oral contraceptives(2 months), serotonin selective reuptake inhibitors (SSRI) (2 weeks), serotonin norepinephrine reuptake inhibitors (SNRI),( 2 weeks) gabapentin, pregabalin, clonidine, selective estrogen receptor modulators, aromatase inhibitors, tissue selective estrogen complexes;(2months)
4. use of aspirin and non-steroidal anti-inflammatory medications for 3 days prior to the SGB procedure; all other anti-platelet or anticoagulation medications will be discontinued with the permission of the participant's prescribing physician
5. for cognition testing: conditions or disorders that can affect performance on cognitive tests (e.g., dementia/mild cognitive impairment, Mini-Mental State Exam (MMSE) less than or equal to 27) at baseline; stroke; traumatic brain injury; alcohol/substance use; inability to write, speak, or read in English, English as a second language, participation in other studies involving tests of cognitive abilities,
6. conditions that can affect depressive symptoms (e.g., current diagnosis of major depression, bipolar disorder, or other Axis I Psychiatric disorder); Personal Health Questionnaire Depression Scale (PHQ-8)> 15
7. Exclusion criteria for neuroimaging study: implantable pulse generators for pacemakers, defibrillator devices and most but not all spinal cord stimulators or deep brain stimulator, ferrous-containing metals within the body (e.g., braces, aneurysm clips, shrapnel/retained particles) inability to tolerate small, enclosed spaces without anxiety (e.g. claustrophobia), weight > 300 lbs. unless height is sufficiently high [e.g., + 5'11"] so that waist and shoulder circumference do not prevent her from fitting in the scanner; opted out of cognition study, shift work
8. Exclusion criteria for SKNA study only allergic to adhesive in electrode

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Changes from baseline and intensity of subjective hot flashes (HF) | Up to 24 weeks (6 months) following intervention
  Changes from baseline of paper diary (subjective) measures of frequency and intensity

SECONDARY OUTCOMES:
Changes from baseline of frequency of objective hot flashes | Up to 24 weeks (6 months) following intervention
  Changes from baseline frequency of objective HFs over a 24 hour period using a validated skin conductance monitor at baseline, 12 weeks (3 months) and 24 weeks (6 months)
Composite changes from baseline of scores of neurocognitive measures | Up to 24 weeks (6 months) following intervention
  Composite changes from baseline of scores to include:California Verbal Learning Test (CVLT) List A, List B, Short-Delay Free Recall, Short-Delay Cued Recall, Long Delay Free Recall, Long Delay Cued Recall, Card Rotation Tests, Finding As, Letter, Semantic and Phonemic Fluency, Logical Memory Subtest of Wechsler Memory Scale (WMS-R/LM-R) Part 1 and (WMS-R/LM-R) Part 2, Mini-Mental State Exam (MMSE), Memory Functioning Questionnaire (MFQ),Closing Question at baseline, 12 weeks (3 months) and 24 weeks (6 months)
Composite changes from baseline of scores of measures of mood | Up to 24 weeks (6 months) following intervention
  Composite changes from baseline of scores of mood to include: Beck Anxiety Inventory (BAI) and Center for Epidemiological Studies-Depression (CES-D) at baseline, 12 weeks (3 months) and 24 weeks (6 months)
Composite changes from baseline of scores of measures of quality of life | Up to 24 weeks (6 months) following intervention
  Composite changes from baseline of scores of quality of life measures to include:Female Sexual Distress Scale (FSDS-R), Menopause Quality of Life Questionnaire (MENQUAL), Patient Global Impression of Change (PGIC), Utian Quality of Life Scale (UQOL), Hot Flash Related Daily Interference Scale (HFRDIS), PAIN Intensity and Interference Scale (PEG) Post Injection Questionnaire at baseline, 12 weeks (3 months) and 24 weeks (6 months)
Changes from baseline of scores of measures of sleep | Up to 24 weeks (6 months) following intervention
  Composite changes from baseline of scores of Pittsburgh Sleep Quality Inventory (PSQI) and Insomnia Severity Index (ISI) at baseline, 12 weeks (3 months) and 24 weeks (6 months)
Changes from baseline of actigraph measures of sleep | Up to 24 weeks (6 months) following intervention
  Changes from baseline of actigraph changes in sleep at baseline, 12 weeks (3 months) and 24 weeks (6 months)
Changes from baseline of Skin Sympathetic Nerve Activity (SKNA) | Up to 2 and 4 weeks following intervention
  Changes of recordings of SKNA using an FDA-approved, specially-configured portable device (Biomation ME6000) in a subset of 60 participants
Changes from baseline of Functional MRI | Up to 12 weeks following intervention
  Changes in fmri activity in a subset of 60 participants at baseline and 3 months following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Hogue, MD, Study Chair — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Paul C. Fitzgerald, Chicago, Illinois